CLINICAL TRIAL: NCT00276003
Title: INST Phase II Trial of Gemcitabine and Irinotecan in Patients With Relapsed or Refractory Lymphoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Ian Rabinowitz, MD; Principal Investigator, University of New Mexico - CRTC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0101C
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-12

CONDITIONS: Non-Hodgkin's Lymphoma; Cancer
Keywords: Lymphoma-Non Hodgkins; Phase II; Gemcitabine; Irinotecan
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms | interventions — Gemcitabine; Irinotecan; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine, Irinotecan, Allopurinol. — Gemcitabine - 1000mg/m2; IV; d1, 8; q 21 days Irinotecan - 100mg/m2; IV; d1, 8; q 21 days Allopurinol - 300 mg; PO; day 1-5; 1st cycle

SUMMARY:
Primary objectives

* Assess the response rate in patients with recurrent or refractory B-cell NHL or Hodgkins disease, treated with the combination of the gemcitabine and irinotecan.

Secondary objectives

* Assess progression free survival in these patients treated with this regimen.
* Assess toxicity of this regimen in this group of patients.

DETAILED DESCRIPTION:
The purpose of the study is to see how well patients with relapsed or refractory lymphoma respond to treatment with Gemcitabine and Irinotecan. Patients on this study take part because they have relapsed or refractory lymphoma. Additionally, the study will assess treatment-related side effects and time until disease progression or recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologic diagnosis of non-HIV related B-cell NHL or Hodgkins disease are eligible.
2. Patients should have documented evidence of refractory or relapsed NHL or Hodgkins disease for inclusion.
3. Patient should have received 1 or more prior chemotherapeutic regimens for relapse, and should have completed last course of treatment at least 3 weeks prior to enrollment.
4. The patient must have bidimensionally measurable or evaluable disease.
5. Age > 18 years.
6. ECOG Performance status < 2
7. Informed consent.
8. ANC > 1.5, platelet count > 100K, creatinine< 2.0, bilirubin < 3
9. Female patients must have a negative pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-08; Primary Completion 2005-06 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Assess the response rate in patients with recurrent or refractory B-cell NHL or Hodgkins disease, treated with the combination of the gemcitabine and irinotecan. | 3 years

SECONDARY OUTCOMES:
Assess progression free survival in these patients with this regimen. | 3 years
Assess toxicity of this regimen in this group of patients. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico
Locations (2):
- United States (2):
  - Lovelace Sandia Health Systems Dept of Hematology, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico